CLINICAL TRIAL: NCT07406282
Title: Double-DARE: Analysis of Doublet and Triplet Therapy With Darolutamide and Other Androgen Receptor Pathway Inhibitors in de Novo mHSPC Patients Seen in Urology Clinics in the USA
Brief Title: A Study to Learn About Real-world Utilization and Outcomes of Darolutamide and Other Androgen Receptor Pathway Inhibitors (ARPIs) for Newly Diagnosed Metastatic Hormone-sensitive Prostate Cancer (de Novo mHSPC) in US Urology Clinics
Acronym: Double-DARE
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23094
Record Dates: First submitted 2025-12-14; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms; Metastatic Hormone-Sensitive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Abiraterone Acetate; enzalutamide; apalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Darolutamide + ADT + docetaxel: Patients receiving darolutamide in combination with androgen deprivation therapy with docetaxel
  Interventions: Drug: Darolutamide
- Abiraterone acetate + ADT + docetaxel: Patients receiving abiraterone acetate in combination with androgen deprivation therapy with docetaxel
  Interventions: Drug: Abiraterone acetate
- Enzalutamide + ADT: Patients receiving enzalutamide in combination with androgen deprivation therapy
  Interventions: Drug: Enzalutamide
- Apalutamide + ADT: Patients receiving apalutamide in combination with androgen deprivation therapy
  Interventions: Drug: Apalutamide
- Darolutamide + ADT: Patients receiving darolutamide in combination with androgen deprivation therapy
  Interventions: Drug: Darolutamide
- Abiraterone acetate + ADT: Patients receiving abiraterone acetate in combination with androgen deprivation therapy
  Interventions: Drug: Abiraterone acetate

INTERVENTIONS:
Drug: Darolutamide — Androgen receptor pathway inhibitor for treatment of metastatic hormone-sensitive prostate cancer
  Other Names: Nubeqa
  Groups: Darolutamide + ADT; Darolutamide + ADT + docetaxel
Drug: Abiraterone acetate — Androgen receptor pathway inhibitor for treatment of metastatic hormone-sensitive prostate cancer
  Groups: Abiraterone acetate + ADT; Abiraterone acetate + ADT + docetaxel
Drug: Enzalutamide — Androgen receptor pathway inhibitor for treatment of metastatic hormone-sensitive prostate cancer
  Groups: Enzalutamide + ADT
Drug: Apalutamide — Androgen receptor pathway inhibitor for treatment of metastatic hormone-sensitive prostate cancer
  Groups: Apalutamide + ADT

SUMMARY:
Prostate cancer is the most common non-skin cancer among men in the United States. For some men, the cancer has already spread to other parts of the body at the time of diagnosis; this is called metastatic hormone-sensitive prostate cancer (mHSPC). Treatment for mHSPC has advanced significantly, with new standards of care involving androgen deprivation therapy (ADT) combined with drugs known as androgen receptor pathway inhibitors (ARPIs), sometimes alongside chemotherapy like docetaxel. Darolutamide is an ARPI that is approved by the FDA for treating mHSPC in a "triplet" combination with ADT and docetaxel. It is also used in a "doublet" combination with ADT alone. However, there is limited information on how darolutamide is used in real-world clinical settings for this condition, which creates a gap in knowledge for making treatment decisions. This study aims to fill that gap by analyzing real-world data from electronic medical records. The primary goal is to describe the characteristics of patients with newly diagnosed mHSPC who are treated with darolutamide (either as a doublet or triplet) in urology clinics across the US. The study will also examine drug use patterns and clinical outcomes for these patients. Additionally, the study will explore the characteristics of patients treated with other ARPIs (abiraterone acetate, enzalutamide, and apalutamide) and assess the feasibility of creating matched patient groups for future comparative research. Data will be collected retrospectively from a large network of community urology practices in the US.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with evidence of de novo mHSPC during the study period
* Initiation of ARPI therapy during the patient identification period and within ±90 days from the mHSPC diagnosis
* Age ≥18 years at index date (ARPI initiation for mHSPC)
* Initiation of ADT and/or docetaxel therapy within ±90 days from index date
* At least 90 days of EMR activity prior to the index date
* At least 90 days of EMR activity post-index, unless the patient died earlier.

Exclusion Criteria:

* History of other primary cancers (except non-melanoma skin cancer)
* Use of PARP inhibitors, chemotherapy (other than docetaxel), immunotherapy or radiopharmaceuticals prior to index date
* Evidence of castration resistance (CR) flag in the database any time before the index date or up to 90 days after the de novo mHSPC diagnosis
* Clinical trial participation during the study period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men with de novo metastatic hormone-sensitive prostate cancer initiating androgen receptor pathway inhibitor therapy in US community urology clinics
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Describe baseline demographic of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): age | Baseline
  Age will be documented in years to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline demographic of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): age | Baseline
  Age will be documented in years to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): Concomitant Medication | Baseline
  Number of concomitant medication will be recorded to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): Concomitant Medication | Baseline
  Number of concomitant medication will be recorded to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline demographic of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): ethnicity | Baseline
  Ethnicity will be documented to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline demographic of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): ethnicity | Baseline
  Ethnicity will be documented to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): Charlson Comorbidity Index | Baseline
  The Charlson Comorbidity Index (CCI) (ranging 0 (no comorbid coonditions) to 5 (high comorbidity burden)) will be determined to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): Charlson Comorbidity Index | Baseline
  The Charlson Comorbidity Index (CCI) (ranging 0 (no comorbid coonditions) to 5 (high comorbidity burden)) will be determined to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): Gleason Score | Baseline
  The Gleason Score (primary and secondary cancer cell pattern are graded on a scale from 1 (least aggressive) to 5 (most aggressive)) will be determined to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): Gleason Score | Baseline
  The Gleason Score (primary and secondary cancer cell pattern are graded on a scale from 1 (least aggressive) to 5 (most aggressive)) will be determined to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): PSA | Baseline
  Most recent prostate specific antigen (PSA) value will be recorded to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): PSA | Baseline
  Most recent prostate specific antigen (PSA) value will be recorded to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy): de novo mHSPC Diagnosis | Baseline
  Record of time from de novo mHSPC diagnosis to Index Date to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe baseline clinical characteristics of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy): de novo mHSPC Diagnosis | Baseline
  Record of time from de novo mHSPC diagnosis to Index Date to characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: initial dose | Day 1 - recorded on the index date (date of first evidence of darolutamide initiation/prescription).
  Document initial dose. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: initial dose | Day 1 - recorded on the index date (date of first evidence of darolutamide initiation/prescription).
  Document initial dose. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: dose change | From index date (Day 1) until the date of the first documented darolutamide dose modification, assessed up to 39 months.
  Document dose change. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: dose change | From index date (Day 1) until the date of the first documented darolutamide dose modification, assessed up to 39 months.
  Document dose change. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: treatment interruption | From index date (Day 1) until the date of the first documented darolutamide interruption, assessed up to 39 months.
  Document period of treatment interruption. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics. Interruptions shorter than 60 days will be considered ongoing treatment (i.e., not counted as a discontinuation).
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: treatment interruption | From index date (Day 1) until the date of the first documented darolutamide interruption, assessed up to 39 months.
  Document period of tretament interruption. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics. Interruptions shorter than 60 days will be considered ongoing treatment (i.e., not counted as a discontinuation).
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: treatment discontinuation | From index date until permanent darolutamide discontinuation, assessed up to 39 months.
  Document permanent treatment discontinuation. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: treatment discontinuation | From index date until permanent darolutamide discontinuation, assessed up to 39 months.
  Document permanent treatment discontinuation. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period:switch to another Androgen receptor pathway inhibitor (ARPI) | From the index date until the date of new ARPI initiation, assessed up to 39 months.
  Date of new ARPI initiation after index; if no prior darolutamide discontinuation recorded, use the day prior to the new ARPI start as darolutamide discontinuation. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period:switch to another Androgen receptor pathway inhibitor (ARPI) | From the index date until the date of new ARPI initiation, assessed up to 39 months.
  Date of new ARPI initiation after index; if no prior darolutamide discontinuation recorded, use the day prior to the new ARPI start as darolutamide discontinuation. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe drug utilization patterns of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period:number of docetaxel cycles (if information is available) | Date of first docetaxel infusion that occurs within ±90 days of index through the last documented docetaxel infusion
  Document number of docetaxel cycles. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: adverse events | From index date (Day 1) through 30 days after recorded end-of-darolutamide treatment
  Document adverse events. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: adverse events | From index date (Day 1) through 30 days after recorded end-of-darolutamide treatment
  Document adverse events. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: comorbid conditions not recorded at baseline | From index date (Day 1) through recorded end of darolutamide treatment, up to 39 months.
  Any new comorbid condition documented from the index date (date of first darolutamide/ARPI initiation) through the recorded end-of-darolutamide treatment in the PPS database. Document comorbid conditions. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period:comorbid conditions not recorded at baseline | From index date (Day 1) through recorded end of darolutamide treatment, up to 39 months.
  Any new comorbid condition documented from the index date (date of first darolutamide/ARPI initiation) through the recorded end-of-darolutamide treatment in the PPS database. Document comorbid conditions. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: PSA response ≥90% | Evaluated at 3, 6, and 12 months from the index treatment.
  Document PSA response ≥90%. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period:PSA response ≥90% | Evaluated at 3, 6, and 12 months from the index treatment.
  Document PSA response ≥90%. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: PSA decline to <0.2 ng/mL (undetectable) | Evaluated at 3, 6, and 12 months from the index treatment.
  Document PSA decline to <0.2 ng/mL (undetectable). Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: PSA decline to <0.2 ng/mL (undetectable) | Evaluated at 3, 6, and 12 months from the index treatment.
  Document PSA decline to <0.2 ng/mL (undetectable). Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: initiation of next antineoplastic therapy | From index date (Day 1) until initiation of next antineoplastic therapy, assessed up to 39 months.
  Document date of next antineoplastic therapy. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: initiation of next antineoplastic therapy | From index date (Day 1) until initiation of next antineoplastic therapy, assessed up to 39 months.
  Document date of next antineoplastic therapy. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: radiographic progression to mCRPC | From index date (Day 1) until radiographic progression to mCRPC, assessed up to 39 months.
  Document radiographic progression to mCRPC. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: radiographic progression to mCRPC | From index date (Day 1) until radiographic progression to mCRPC, assessed up to 39 months.
  Document radiographic progression to mCRPC. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT + docetaxel (triplet therapy) during the study period: all-cause mortality | From index date (Day 1) until death from any cause, assessed up to 39 months.
  Date of death. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT + docetaxel in adult men diagnosed with de novo mHSPC in US urology clinics.
Describe treatment outcomes of de novo mHSPC patients receiving darolutamide + ADT (doublet therapy) during the study period: all-cause mortality | From index date (Day 1) until death from any cause, assessed up to 39 months.
  Date of death. Characterize the real-world utilization and treatment outcomes for the darolutamide combination with ADT in adult men diagnosed with de novo mHSPC in US urology clinics.

CONTACTS AND LOCATIONS:
Locations (1):
- Precision Point Specialty LLC PPS Analytics, a Specialty Networks LLC Company, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No